CLINICAL TRIAL: NCT05845008
Title: An Open-label, Single-arm, Multiple-dose Study to Evaluate the Safety of a Fixed Combination of Acetaminophen/Naproxen Sodium in Adolescents 12 to Less Than 17 Years of Age With Orthodontic Pain
Brief Title: A Multiple-Dose Safety Study of Fixed Combination of Acetaminophen/Naproxen Sodium in Adolescents With Orthodontic Pain
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study is no longer required due to change in development program strategy.
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCSPAP005204; CCSPAP005204 (Other: Johnson & Johnson Consumer Inc. (J&JCI))
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Orthodontic Pain
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Acetaminophen/Naproxen Sodium Fixed Combination (Experimental): Participants will self-administer a fixed combination of acetaminophen/naproxen sodium orally as multiple doses over a period of up to 10 days.
  Interventions: Drug: Acetaminophen/Naproxen Sodium Fixed Combination

INTERVENTIONS:
Drug: Acetaminophen/Naproxen Sodium Fixed Combination — Acetaminophen/naproxen sodium fixed combination tablets, oral.

SUMMARY:
The purpose of this study is to evaluate the safety of a fixed combination of acetaminophen/naproxen sodium when administered as multiple doses over a period of up to 10 days in adolescents 12 to below 17 years of age with post-procedure orthodontic pain.

ELIGIBILITY:
Inclusion Criteria:

* Weigh 72 pounds or greater and have a body mass index (BMI)-for-age between the 5th and 95th percentile (inclusive) at Screening
* Have undergone an orthodontic procedure within 4 hours prior to baseline (enrollment) visit
* Females of childbearing potential and males agree to the contraceptive requirements of study

Exclusion Criteria:

* Are female and are pregnant, breastfeeding, or trying to become pregnant or male with a pregnant partner or a partner currently trying to become pregnant
* Have a positive urine drug test on screening or enrollment
* Are not able to swallow whole tablets or capsules
* Arrive at the site on the day of enrollment with motion sickness and/or have a history of frequent motion sickness (car sickness) in the past year, which in the judgement of the investigator is likely to confound assessment of adverse events
* Routinely use oral analgesics greater than or equal to (>=) 5 times per week
* Have a known allergy or hypersensitivity to naproxen (or other nonsteroidal anti-inflammatory drugs including aspirin) or acetaminophen or have asthma
* Have presence or a history of major medical condition that in the Investigator's opinion may jeopardize the participant's safety or wellbeing or the integrity of the study
* Have a history of chronic use of tranquilizers, alcohol, tobacco/vaping, or substance abuse, as judged by the Investigator site staff, in the last year
* Have a history of endoscopically documented peptic ulcer disease or bleeding disorder in the last two years
* Have a diagnosis of gastroesophageal reflux disorder, or experienced frequent heartburn in the past year

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-07-26 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to Day 10
  An adverse event (AE) is any untoward medical occurrence that occurs in a participant after he/she has signed an informed consent for a study. The event does not need to have a suspected causal relationship with the investigational product (IP). A TEAE is an AE that occurs after the first dose of study drug, or an AE that started before the first use of study drug and worsened after taking the study drug.
Number of Participants with Serious Adverse Events (SAEs) | Up to Day 10
  An AE is any untoward medical occurrence that occurs in a participant after he/she has signed an informed consent for a study. The event does not need to have a suspected causal relationship with the IP. A SAE is an AE or suspected adverse reaction resulting in any of the following outcomes: result in death; is life-threatening (immediate risk of death); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions; results in congenital anomaly/birth defect; is considered medically significant; is a suspected transmission of any infectious agent via a medical product.
Number of Participants with Treatment-related AEs | Up to Day 10
  An AE is any untoward medical occurrence that occurs in a participant after he/she has signed an informed consent for a study. The event does not need to have a suspected causal relationship with the IP. Treatment-related AEs are adverse events evaluated by the investigator as possible, probable or very likely related to investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Bertoch, Principal Investigator — JBR Clinical Research
Locations (1):
- JBR Clinical Research LLP, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu